CLINICAL TRIAL: NCT04097379
Title: A Randomized, Placebo-controlled, Subject and Investigator Blinded Study Investigating the Safety, Tolerability and Preliminary Efficacy of 8-week Treatment With Intra-articular LRX712 to Regenerate Articular Cartilage in Patients With Mild/Moderate Knee Osteoarthritis
Brief Title: Safety, Tolerability and Preliminary Efficacy of Multiple Intra-articular Injections of LRX712 in Patients With Knee OA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLRX712A12201; 2019-002963-92 (EudraCT Number)
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis (OA)
Keywords: Knee osteoarthritis; Chondroanabolic drug; Magnetic resonance imaging; Patient Reported Outcomes
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LRX712 15 mg (Experimental): LRX712 15 mg was administered intra-articularly (i.a.) every four weeks, for a total of three administrations.
  Interventions: Drug: LRX712
- LRX712 25 mg (Experimental): LRX712 25 mg was administered i.a. every four weeks, for a total of three administrations.
  Interventions: Drug: LRX712
- LRX712 75 mg (Experimental): LRX712 75 mg was administered i.a. every four weeks, for a total of three administrations.
  Interventions: Drug: LRX712
- Placebo (Placebo Comparator): Placebo was administered i.a. every four weeks, for a total of three administrations.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LRX712 — LRX712 intra-articular injections
  Arms: LRX712 15 mg; LRX712 25 mg; LRX712 75 mg
Other: Placebo — Placebo intra-articular injections
  Arms: Placebo

SUMMARY:
This study explored the preliminary efficacy of multiple intra-articular injections of LRX712 by evaluating the ability of the drug to restore structural integrity of articular cartilage. Efficacy was evaluated in the context of the systemic safety and local tolerability of the investigational drug.

DETAILED DESCRIPTION:
This was an exploratory study, with a 7-week screening period, an 8-week treatment period, and a 44-week follow-up period, using a 3-treatment arm, parallel-group, randomized, double-blind, placebo-controlled clinical study design. The study design implemented for the first six participants enrolled was a 2-treatment arm, parallel -group, randomized, double-blind placebo controlled trial (up until the time when the study was temporarily halted in February 2021) included up to 5 weeks of screening, an 8-week treatment period, and a 44-week follow-up period. The original two-arm study design (75 mg LRX712 vs. placebo) was modified to a three-arm design, with two lower doses of LRX712 (15 mg and 25 mg) vs. placebo, following protocol amendment 4 (16-Jul-2021). Data from the three participants who had completed dosing with 75 mg LRX712 were considered exploratory, and data from the three participants who had completed dosing with placebo were pooled with the data from participants enrolled after the study was restarted with the implementation of protocol amendment 4.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained before any assessment is performed.

To be eligible for inclusion in this study patients must meet all of the following criteria:

* Patient must have a BMI between 18 -35 kg/m2
* Patient must have symptomatic knee osteoarthritis predominantly in one knee (index knee)
* Patient must have knee osteoarthritis (Kellgren-Lawrence grade 2 or 3) in the index knee, as confirmed by radiography
* Patient must have radiographic confirmation of a medial joint space width of 1.5 to 3.5 mm for females, or 2 to 4 mm for males within the medial tibio-femoral compartment of the index knee.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for inclusion in this study:

* Patient has a known autoimmune disease, inflammatory or chronic arthropathy other than OA.
* Patient had partial or complete joint replacement in one or both knees.
* Patient has symptomatic, isolated patello-femoral pain in the index knee as per the Investigator's examination.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Previous use of LRX712 or use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations.
* Patient has malalignment (valgus- or varus-deformity) ≥ 7.5° in the index knee as per anatomic PA axis measured by weight-bearing short knee radiography.
* History of significant cardiac conduction/electrophysiological disorder, e.g. familial long QT syndrome or known family history of Torsades de Pointes or prolonged QT syndrome or QTcF ≥ 450 msec (Fridericia Correction) for males and ≥ 460 msec for females at screening or baseline (by local 12-lead digitized ECG reading).
* Signs or symptoms, in the judgment of the investigator, of a clinically significant systemic viral, bacterial or fungal infection within 30 days prior to screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 1 investigative site in Netherlands.
Pre-assignment Details: This study had a 7-week screening period.
Period: Overall Study
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg | Placebo
Started | 12 | 14 | 3 | 16
Completed | 11 | 13 | 3 | 16
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg | Placebo | Total
Number analyzed (Participants) | 12 | 14 | 3 | 16 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.74) | 61.6 (7.31) | 59.7 (5.03) | 58.4 (8.66) | 61.6 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 1 | 7 | 20
  Male | 7 | 7 | 2 | 9 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 0 | 2
  White | 11 | 13 | 3 | 16 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cartilage Volume in the Index Region Measured by 7 Tesla MRI
Description: Magnetic resonance images (MRI) were obtained from the target knee to visualize and quantify changes in the volume of cartilage in the index region. The index region was defined as the combination of the femoral medial anterior (FMA), central (FMC) and posterior (FMP) cartilage subregions in the knee. Change from baseline in cartilage volume was analyzed using the mixed effects model for repeated measures (MMRM). The model included baseline, treatment, timepoint and treatment-timepoints as fixed effects, and participant as random effect. Missing data was assumed to be Missing at Random (MAR).
Time Frame: Baseline, Week 28
Population: Participants in the safety analysis set from the arms "LRX712 15 mg", "LRX712 25 mg" and "Placebo" who had an available value for the outcome measure as aligned with protocol. The Safety Set comprises all enrolled participants who received any investigational treatment.
Measure: Least Squares Mean (Standard Error); unit: µL
Arm/Group | LRX712 15 mg | LRX712 25 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 16
µL | 63.3 (54.93) | 49.8 (50.57) | 11.6 (45.54)
Statistical Analysis 1: Comparison: LRX712 15 mg vs Placebo; Test type: Superiority; p = 0.2366, Mixed effects model for repeated measure; Least Square Mean = 51.70, 90% CI [-68.7 to 172.1], Standard Error of Mean 71.327
Statistical Analysis 2: Comparison: LRX712 25 mg vs Placebo; Test type: Superiority; p = 0.2892, Mixed effects model for repeated measure; Least Square Mean = 38.19, 90% CI 2-sided [-76.7 to 153.1], Standard Error of Mean 68.100

2. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of LRX712
Description: Tmax is the time to reach maximum (peak) LRX712 concentration after single-dose administration (time). LRX712 plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). LRX712 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 25 pg/mL.
Time Frame: Pre-dose, 0.5, 12, 24 and 168 hours after dose on Day 1; Pre-dose, 24 and 168 hours after dose on Day 29; Pre-dose, 24, 168, 1344 and 3360 hours after dose on Day 57
Population: Pharmacokinetic (PK) analysis set: Includes all participants with at least one available valid PK concentration measurement, who received any dose of LRX712 and with no protocol deviations that impact on PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 12 | 14 | 3
hours
  Day 1 | 17.5 [12.0 to 24.0] | 23.3 [0.50 to 24.1] | 24.0 [12.0 to 24.1]
  Day 29: number analyzed (Participants) | 10 | 13 | 2
  Day 29 | 23.8 [22.6 to 24.0] | 24.0 [22.2 to 24.2] | 23.9 [23.8 to 24.0]
  Day 57: number analyzed (Participants) | 11 | 13 | 3
  Day 57 | 24.0 [21.9 to 24.0] | 24.0 [22.0 to 24.1] | 24.0 [23.5 to 24.0]

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of LRX712
Description: Cmax is defined as the maximum (peak) observed concentration following a dose. LRX712 plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). LRX712 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 25 pg/mL.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 12 | 14 | 3
ng/mL
  Day 1 | 3.52 (2.07) | 6.54 (5.33) | 6.94 (4.96)
  Day 29: number analyzed (Participants) | 10 | 13 | 2
  Day 29 | 3.33 (2.57) | 3.50 (1.43) | 27.0 (31.6)
  Day 57: number analyzed (Participants) | 11 | 13 | 3
  Day 57 | 2.39 (0.951) | 4.05 (2.25) | 29.5 (20.4)

4. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of LRX712
Description: Cmin is defined as the minimum (peak) observed concentration following a dose. LRX712 plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). LRX712 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 25 pg/mL.
Time Frame: Pre-dose on Day 29; Pre-dose, 1344 hours after dose on Day 57 (LRX712 15 mg arm) and 3360 hours after dose on Day 57 (LRX712 25 mg and 75 mg arms)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 11 | 14 | 3
ng/mL
  Dose 1 (pre-dose Day 29): number analyzed (Participants) | 10 | 14 | 3
  Dose 1 (pre-dose Day 29) | 0.0735 (0.10) | 0.0823 (0.115) | 0.231 (0.401)
  Dose 2 (pre-dose Day 57): number analyzed (Participants) | 11 | 13 | 3
  Dose 2 (pre-dose Day 57) | 0.111 (0.109) | 0.202 (0.204) | 0.365 (0.585)
  Dose 3 (post-dose Day 57): number analyzed (Participants) | 10 | 12 | 3
  Dose 3 (post-dose Day 57) | 0.0439 (0.0740) | 0.00379 (0.0131) | 0.0120 (0.0208)

5. Secondary Outcome: Synovial Fluid Concentrations of LRX712
Description: The observed synovial concentration following a dose. LRX712 concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). LRX712 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 20 ng/mL. Samples were collected from a limited number of participants.
Time Frame: Pre-dose on Day 1, 29 and 57
Population: Participants in the PK analysis set with a synovial sample collected and a valid value for the outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 2 | 3 | 0
ng/mL
  Day 1: number analyzed (Participants) | 1 | 2 | 0
  Day 1 | 0 | 0 (0) |
  Day 29: number analyzed (Participants) | 1 | 1 | 0
  Day 29 | 0 | 0 |
  Day 57: number analyzed (Participants) | 0 | 2 | 0
  Day 57 |  | 0 (0) |

6. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of MAE344
Description: Tmax is the time to reach maximum (peak) MAE344 concentration after single-dose administration (time). MAE344 is a metabolite of LRX712 and plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). MAE344 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 100 pg/mL.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 12 | 14 | 3
hours
  Day 1 | 23.5 [12.0 to 24.1] | 24.0 [12.0 to 169] | 24.1 [24.0 to 24.1]
  Day 29: number analyzed (Participants) | 10 | 13 | 2
  Day 29 | 23.8 [22.6 to 24.0] | 24.0 [22.2 to 193] | 23.9 [23.8 to 24.0]
  Day 57: number analyzed (Participants) | 11 | 13 | 3
  Day 57 | 24.0 [21.9 to 169] | 24.0 [22.0 to 24.1] | 24.0 [23.5 to 24.0]

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MAE344
Description: Cmax is defined as the maximum (peak) observed concentration following a dose. MAE344 is a metabolite of LRX712 and plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). MAE344 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 100 pg/mL.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 12 | 14 | 3
ng/mL
  Day 1 | 38.3 (23.0) | 52.1 (47.3) | 75.2 (63.1)
  Day 29: number analyzed (Participants) | 10 | 13 | 2
  Day 29 | 42.6 (37.4) | 40.5 (24.6) | 281 (329)
  Day 57: number analyzed (Participants) | 11 | 13 | 3
  Day 57 | 26.0 (11.8) | 45.1 (33.7) | 321 (170)

8. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of MAE344
Description: Cmin is defined as the minimum (peak) observed concentration following a dose. MAE344 is a metabolite of LRX712 and plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). MAE344 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 100 pg/mL.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 11 | 14 | 3
ng/mL
  Dose 1 (pre-dose Day 29): number analyzed (Participants) | 10 | 14 | 3
  Dose 1 (pre-dose Day 29) | 1.34 (1.76) | 1.49 (1.82) | 4.11 (7.01)
  Dose 2 (pre-dose Day 57): number analyzed (Participants) | 11 | 13 | 3
  Dose 2 (pre-dose Day 57) | 2.12 (2.15) | 3.04 (3.06) | 5.70 (9.10)
  Dose 3 (post-dose Day 57): number analyzed (Participants) | 10 | 12 | 3
  Dose 3 (post-dose Day 57) | 0.916 (1.22) | 0.0557 (0.140) | 0.257 (0.445)

9. Secondary Outcome: Synovial Fluid Concentrations of MAE344
Description: The observed synovial concentration following a dose. MAE344 is a metabolite of LRX712 and concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). MAE344 was determined by a validated LC-MS/MS method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero" . LLOQ was 80 ng/mL. Samples were collected from a limited number of participants.
Time Frame: Pre-dose on Day 1, 29 and 57
Population: Participants in the PK analysis set with a synovial sample collected and a valid value for the outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg
Number analyzed (Participants) | 2 | 3 | 0
ng/mL
  Day 1: number analyzed (Participants) | 1 | 2 | 0
  Day 1 | 0 | 0 (0) |
  Day 29: number analyzed (Participants) | 1 | 1 | 0
  Day 29 | 0 | 0 |
  Day 57: number analyzed (Participants) | 0 | 2 | 0
  Day 57 |  | 0 (0) |

10. Secondary Outcome: Change From Baseline in Articular Cartilage [23Na] Content Measured by 7 Tesla MRI
Description: Magnetic resonance images (MRI) were obtained from the target knee to visualize and quantify changes in articular cartilage quality (assessed by changes in glycosaminoglycans content measured by sodium content) in the index region. The index region was defined as the combination of the femoral medial anterior (FMA), central (FMC) and posterior (FMP) cartilage subregions in the knee quality. Change from baseline in articular cartilage content was analyzed using a mixed effects model for repeated measures (MMRM). The model included baseline, treatment, timepoint and treatment-timepoints as fixed effects, and participant as random effect. Missing data was assumed to be Missing at Random (MAR). The data from the three participants who completed dosing with 75 mg LRX712 were considered exploratory.
Time Frame: Baseline, Week 16, 28 and 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | LRX712 15 mg | LRX712 25 mg | Placebo
Number analyzed (Participants) | 9 | 11 | 16
mmol/L
  Week 16: number analyzed (Participants) | 8 | 8 | 14
  Week 16 | -7.4 (12.00) | 12.7 (11.99) | 8.5 (9.20)
  Week 28: number analyzed (Participants) | 9 | 9 | 13
  Week 28 | -15.5 (11.21) | 8.9 (11.13) | 4.0 (9.24)
  Week 52 | 3.1 (12.12) | 26.6 (11.19) | 5.5 (9.20)

11. Secondary Outcome: Change From Baseline in Cartilage Volume in the Index Region Measured by 7 Tesla MRI
Description: Magnetic resonance images (MRI) were obtained from the target knee to visualize and quantify changes in volume of cartilage in the index region. The index region was defined as the combination of the femoral medial anterior (FMA), central (FMC) and posterior (FMP) cartilage subregions in the knee quality. Change from baseline in cartilage volume was analyzed using a mixed effects model for repeated measures (MMRM). The model included baseline, treatment, timepoint and treatment-timepoints as fixed effects, and participant as random effect. Missing data was assumed to be Missing at Random (MAR). The data from the three participants who completed dosing with 75 mg LRX712 were considered exploratory.
Time Frame: Baseline, Week 16 and 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µL
Arm/Group | LRX712 15 mg | LRX712 25 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 16
µL
  Week 16: number analyzed (Participants) | 10 | 11 | 15
  Week 16 | -48.0 (52.64) | -17.4 (50.09) | 24.4 (43.05)
  Week 52 | 19.5 (73.11) | 49.3 (67.29) | 123.1 (60.62)

ADVERSE EVENTS:
Time Frame: Adverse events were reported as "on-treatment" from first dose until last dose of study treatment plus 30 days and as "follow up" from last dose of study treatment plus 29 days up to a maximum duration of approximately 52 weeks.
Groups:
- LRX712 15mg and 25mg; LRX712 15mg and 25mg_Post-treatment: LRX712 was administered i.a. every four weeks, for a total of three administrations.
- LRX712 15 mg_Post-treatment: LRX712 15 mg was administered intra-articularly (i.a.) every four weeks, for a total of three administrations.
- LRX712 25 mg_Post-treatment: LRX712 25 mg was administered i.a. every four weeks, for a total of three administrations.
- LRX712 75 mg_Post-treatment: LRX712 75 mg was administered i.a. every four weeks, for a total of three administrations.
- Placebo_Post-treatment: Placebo was administered i.a. every four weeks, for a total of three administrations.
- Total: Total
Arm/Group | LRX712 15 mg | LRX712 25 mg | LRX712 75 mg | LRX712 15mg and 25mg | Placebo | LRX712 15 mg_Post-treatment | LRX712 25 mg_Post-treatment | LRX712 75 mg_Post-treatment | LRX712 15mg and 25mg_Post-treatment | Placebo_Post-treatment | Total
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/3 | 0/26 | 0/16 | 0/12 | 0/14 | 0/3 | 0/26 | 0/16 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/3 | 0/26 | 0/16 | 1/12 | 1/14 | 0/3 | 2/26 | 1/16 | 3/45
Other Adverse Events (participants affected / at risk) | 11/12 | 14/14 | 3/3 | 25/26 | 16/16 | 7/12 | 7/14 | 0/3 | 14/26 | 13/16 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LRX712 15 mg (N=12) | LRX712 25 mg (N=14) | LRX712 75 mg (N=3) | LRX712 15mg and 25mg (N=26) | Placebo (N=16) | LRX712 15 mg_Post-treatment (N=12) | LRX712 25 mg_Post-treatment (N=14) | LRX712 75 mg_Post-treatment (N=3) | LRX712 15mg and 25mg_Post-treatment (N=26) | Placebo_Post-treatment (N=16) | Total (N=45)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LRX712 15 mg (N=12) | LRX712 25 mg (N=14) | LRX712 75 mg (N=3) | LRX712 15mg and 25mg (N=26) | Placebo (N=16) | LRX712 15 mg_Post-treatment (N=12) | LRX712 25 mg_Post-treatment (N=14) | LRX712 75 mg_Post-treatment (N=3) | LRX712 15mg and 25mg_Post-treatment (N=26) | Placebo_Post-treatment (N=16) | Total (N=45)
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 4
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 2 | 1 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 10
Malaise (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 5
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 7 | 4 | 3 | 2 | 0 | 5 | 4 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 | 7 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 8 | 1 | 13 | 12 | 0 | 1 | 0 | 1 | 2 | 27
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT04097379/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT04097379/SAP_001.pdf